CLINICAL TRIAL: NCT07213232
Title: Investigation of the Effects of Dual-Task Balance and Gait Training Combined With Cognitive Training in Parkinson's Patients
Brief Title: Dual-Task Balance and Gait Training Combined With Cognitive Training in Parkinson's Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: T.C. Sağlık Bakanlığı Ankara Bilkent Şehir Hastanesi (Other)
Responsible Party: Principal Investigator, Arzu Güçlü Gündüz, Professor, PhD, PT, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TABED 1/ 985/ 2025
Record Dates: First submitted 2025-09-19; First posted 2025-10-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cognition; Parkinson's Disease; Gait Disorders, Neurologic; Balance Disorders
Keywords: dual-task training; cognitive training; balance; gait; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training Combined with Dual-Task Training Group (DUAL-COG) (Experimental): The intervention will start with core stability training, followed by dual-task balance and gait training. After completion of the dual-task training phase, participants will undergo structured cognitive training.
  Interventions: Other: Core Stability Training; Other: Dual-Task Balance and Gait Training; Other: Cognitive Training
- Dual-Task Training Group (DUAL) (Active Comparator): The intervention will start with core stability training, followed by dual-task balance and gait training.
  Interventions: Other: Core Stability Training; Other: Dual-Task Balance and Gait Training

INTERVENTIONS:
Other: Core Stability Training — Core stability training will be designed to prepare participants for subsequent balance and gait exercises by promoting normal proprioceptive input through activation of deep core muscles. This training will be performed in the supine position at the beginning of each session for both groups.
Other: Dual-Task Balance and Gait Training — Dual-task balance and gait training will be provided with task-oriented motor-cognitive and motor-motor exercises with the augmented and virtual reality system C-Mill VR+ (Motek Medical, Amsterdam, The Netherlands). Sessions will be individualized based on each participant's current abilities and the difficulty level of the tasks to address specific patient needs. Each training session will have a duration of 30 minutes for both groups.
Other: Cognitive Training — Cognitive training will be provided with RehaCom software, a program that emphasizes learning principles, provides task-specific exercises, delivers positive feedback, and allows individualized progression based on patient-specific difficulty levels. In the present study, the cognitive training will target the "Attention," "Memory," and "Executive Functions" domains, which are known to be affected from the early stages of Parkinson's disease. Exercises will be initiated at a level appropriate to each participant's cognitive abilities and will gradually increase in difficulty. Each training session will have a duration of 30 minutes.
  Arms: Cognitive Training Combined with Dual-Task Training Group (DUAL-COG)

SUMMARY:
The aim of the study is to examine the effects of a structured, cognitive dimension-specific cognitive training combined with dual-task balance and gait training on balance, gait, and cognition in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the most common movement disorder and the second most prevalent neurodegenerative disease after Alzheimer's disease. In addition to cardinal motor symptoms such as bradykinesia, rigidity, and resting tremor, PD is associated with a wide spectrum of non-motor symptoms that substantially increase overall disease burden. Among these, cognitive impairment is particularly significant, occurring up to six times more frequently in individuals with PD compared to the healthy population.

Although research on cognition in PD has increased over the past two decades, knowledge and treatment strategies for cognitive deficits remain limited compared to those addressing motor symptoms. Since no effective treatment currently exists to prevent or delay cognitive decline in PD, investigations into cognitive interventions are gaining increasing importance for understanding and managing this disabling aspect of the disease, which may emerge at all stages.

One promising intervention is RehaCom, a computer-based program that provides personalized cognitive training modules tailored to individual needs. Previous studies have demonstrated that RehaCom improves cognitive performance, enhances quality of life, and optimizes function in impaired domains. By prioritizing learning principles and offering individualized training for specific cognitive dimensions, RehaCom has also been shown to promote neural plasticity in patients with PD.

Motor learning literature emphasizes that not only training intensity but also conditions resembling real-life scenarios are critical for effective rehabilitation. Daily activities often require walking and maintaining balance while simultaneously performing additional tasks, such as speaking (cognitive dual-task) or carrying an object (motor dual-task). Dual-task training, which integrates motor training with either a cognitive or an additional motor task, is a comprehensive approach supported by strong evidence. Compared to single-task practice, dual-task training enhances motor learning, yields greater functional gains, and facilitates transfer of these improvements to activities of daily living.

Considering the deficiencies in cognition as a reason for the progressive and irreversible nature of the pathogenesis of PD, the present study hypothesizes that providing structured cognitive skills training will be more effective in improving both motor and cognitive functions. However, a review of the literature indicates that studies in this area remain limited. Therefore, the present study aims to implement and evaluate a rehabilitation program combining cognitive training with dual-task-focused balance and gait exercises in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with idiopathic Parkinson's disease by a neurologist.
* Evaluated between Stage 1-3 according to the Hoehn and Yahr Staging Scale.
* Aged 40 years or older.
* Agreed to participate in the study after being given sufficient information.

Exclusion Criteria:

* Patients with a Montreal Cognitive Assessment score of 20 and below.
* Patients with cardiovascular, vestibular, musculoskeletal or additional neurological disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Static Standing Balance Parameters at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The static standing balance of participants will be assessed using the Huber 360° Evolution System (LPG Systems, Valence, France). The following measurements will be performed with this device:
  Postural Stability Test: Postural stability will be evaluated in parallel feet (eyes open/closed) and single-leg positions. Each test will be repeated three times, with a 10-second rest interval between repetitions. The displacement area (mm²), and path length (mm) of the center of pressure will be recorded. Additionally, during the test, the displacement of the center of pressure per unit time will be recorded as velocity (mm/s).
Change from Baseline in Dynamic Standing Balance Parameters at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The dynamic standing balance of participants will be assessed using the Huber 360° Evolution System (LPG Systems, Valence, France). The following measurements will be performed with this device:
  Limits of Stability Test: During the test, participants will be instructed to shift their weight toward eight different directions. Each test will be repeated three times, with a 10-second rest interval between repetitions. Outcome measures will include the displacement of the center of pressure in each direction (mm) and the sway area (mm²) resulting from the displacement of the center of pressure across all directions.
Change from Baseline in Spatial Gait Analysis Parameters at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The C-Mill VR+ system (Motek Medical, Amsterdam, The Netherlands) will be used for the evaluation. The analysis will include the recording of step length (mm), step width (mm) and stride length (mm).
Change from Baseline in Temporal Gait Analysis Parameters at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The C-Mill VR+ system (Motek Medical, Amsterdam, The Netherlands) will be used for the evaluation. The analysis will include the recording of stance phase duration (ms), swing phase duration (ms), and double support phase duration (ms).
Change from Baseline in Walking Distance Parameter at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The C-Mill VR+ system (Motek Medical, Amsterdam, The Netherlands) will be used for the evaluation. The analysis will include the recording of walking distance (m) as a functional performance outcome.
Change from Baseline in Gait Speed at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The C-Mill VR+ system (Motek Medical, Amsterdam, The Netherlands) will be used in the evaluation. The analysis will include recording the displacement of the individual per unit time on the running belt as gait speed (m/s).
Change from Baseline in Montreal Cognitive Assessment (MoCA) Score at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  Montreal Cognitive Assessment (MoCA), which provides a general cognitive screening in different cognitive functions such as attention, concentration, executive functions, memory, language, visual structuring skills, abstract thought, calculation and orientation, will be used in the general evaluation of cognition. MoCA is an effective scale especially in the evaluation of mild cognitive impairments in Parkinson's disease (PD). The cut-off score range of MoCA has been shown to be 18-26 points in individuals with PD who has mild cognitive impairment. The administration of MoCA takes approximately 10 minutes. The highest total score that can be obtained from the test is 30. Accordingly, a score of 21 points and above is considered normal.
Change in Domain-Specific Cognitive Assessment Parameters from Baseline after 12 Training Sessions | From enrollment to the end of the 6-Week training program
  In the comprehensive evaluation of cognition, specific evaluation will be made for the sub-domains of cognition which are "Attention", "Memory" and "Executive Functions" will be made using the screening modules of the RehaCom software. Before each evaluation, a practice mode will be applied in which the patient is informed about the things to be careful about during the evaluation, the expected task and the purpose of the evaluation. In all screening results, the z-values, mean of reaction time (ms), median of reaction time (ms), standard deviation of reaction time (ms) and correct, incorrect, error and skip numbers in the tests will be recorded as standardized data compared with the data of at least 200 age and gender matched healthy individuals in RehaCom's database.

SECONDARY OUTCOMES:
Change from Baseline in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3: Motor Examination Scores at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) consists of 4 parts, like the classic UPDRS. The severity of the patients' motor symptoms will be assessed using the Motor Examination part, which is the 3rd part of the MDS-UPDRS. MDS-UPDRS Part 3 consists of 18 items. All items in the scale are scored between 0 (Normal) and 4 (Severe) points.
Change from Baseline in Activities-Specific Balance Confidence (ABC) Scale Scores at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  The level of confidence felt by the patient in daily life activities requiring balance skills will be evaluated with the Activities-Specific Balance Confidence (ABC) Scale. In this scale, individuals are asked to rate the sense of security they feel while performing 16 activities requiring balance skills between 0% and 100%.
Change from Baseline in Percentile of Evaluation of Dual-Task Effect at 12 Training Sessions | From enrollment to the end of the 6-Week training program
  In addition to gait speed, the effect of dual-task on gait speed will be assessed by calculating the dual-task cost using the following formula:
  [(Dual Task Gait Speed-Single Task Gait Speed)/(Single Task Walking Speed)] x 100%

CONTACTS AND LOCATIONS:
Overall Officials: Emre Adıgüzel, Prof., MD., Study Director — Ankara Bilkent City Hospital Physical Medicine and Rehabilitation Hospital; Arzu Güçlü Gündüz, Prof., PT., Study Director — Gazi University
Locations (1):
- Ankara Bilkent City Hospital Physical Medicine and Rehabilitation Hospital, Ankara, Üniversiteler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernini S, Alloni A, Panzarasa S, Picascia M, Quaglini S, Tassorelli C, Sinforiani E. A computer-based cognitive training in Mild Cognitive Impairment in Parkinson's Disease. NeuroRehabilitation. 2019;44(4):555-567. doi: 10.3233/NRE-192714. PMID 31256092
- [Background] Yogev G, Giladi N, Peretz C, Springer S, Simon ES, Hausdorff JM. Dual tasking, gait rhythmicity, and Parkinson's disease: which aspects of gait are attention demanding? Eur J Neurosci. 2005 Sep;22(5):1248-56. doi: 10.1111/j.1460-9568.2005.04298.x. PMID 16176368
- [Background] Rochester L, Hetherington V, Jones D, Nieuwboer A, Willems AM, Kwakkel G, Van Wegen E. Attending to the task: interference effects of functional tasks on walking in Parkinson's disease and the roles of cognition, depression, fatigue, and balance. Arch Phys Med Rehabil. 2004 Oct;85(10):1578-85. doi: 10.1016/j.apmr.2004.01.025. PMID 15468014
- [Background] Fritz NE, Cheek FM, Nichols-Larsen DS. Motor-Cognitive Dual-Task Training in Persons With Neurologic Disorders: A Systematic Review. J Neurol Phys Ther. 2015 Jul;39(3):142-53. doi: 10.1097/NPT.0000000000000090. PMID 26079569
- [Background] Cerasa A, Gioia MC, Salsone M, Donzuso G, Chiriaco C, Realmuto S, Nicoletti A, Bellavia G, Banco A, D'amelio M, Zappia M, Quattrone A. Neurofunctional correlates of attention rehabilitation in Parkinson's disease: an explorative study. Neurol Sci. 2014 Aug;35(8):1173-80. doi: 10.1007/s10072-014-1666-z. Epub 2014 Feb 20. PMID 24554416
- [Background] Leung IH, Walton CC, Hallock H, Lewis SJ, Valenzuela M, Lampit A. Cognitive training in Parkinson disease: A systematic review and meta-analysis. Neurology. 2015 Nov 24;85(21):1843-51. doi: 10.1212/WNL.0000000000002145. Epub 2015 Oct 30. PMID 26519540
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886
- [Background] Aarsland D, Andersen K, Larsen JP, Lolk A, Nielsen H, Kragh-Sorensen P. Risk of dementia in Parkinson's disease: a community-based, prospective study. Neurology. 2001 Mar 27;56(6):730-6. doi: 10.1212/wnl.56.6.730. PMID 11274306
- [Background] Zaman V, Shields DC, Shams R, Drasites KP, Matzelle D, Haque A, Banik NL. Cellular and molecular pathophysiology in the progression of Parkinson's disease. Metab Brain Dis. 2021 Jun;36(5):815-827. doi: 10.1007/s11011-021-00689-5. Epub 2021 Feb 18. PMID 33599945